CLINICAL TRIAL: NCT00719160
Title: Dietary Protein's Effect on Gastric pH and Calcium Absorption
Brief Title: The Effect of Protein on Calcium Absorption and Gastric Acid Production
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0910005852; 129772 (Other Grant/Funding Number: Other Federal ID)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Osteoporosis
Keywords: Gastric acid; Dietary protein; Calcium; Intestinal absorption; Calcium sensing receptor
MeSH Terms: conditions — Osteoporosis | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esomeprazole (Placebo Comparator)
  Interventions: Drug: esomeprazole; Drug: Placebo
- Placebo (Active Comparator)
  Interventions: Drug: esomeprazole; Drug: Placebo

INTERVENTIONS:
Drug: esomeprazole — 2 Interventions with esomeprazole 20 mg twice a day for 9 days vs. a placebo for 9 days while on a high protein diet
Drug: Placebo — Placebo 20 mg twice a day for 9 days

SUMMARY:
We have established that dietary protein is an important regulator of intestinal calcium absorption in humans. However, we do not understand the mechanism by which dietary protein is affecting calcium absorption. Therefore, the purpose of this research is to evaluate whether dietary protein-induced changes in gastric acid secretion explain the observed changes in intestinal calcium absorption.

DETAILED DESCRIPTION:
We have established that dietary protein is an important regulator of intestinal calcium absorption in humans. However, we do not understand the mechanism by which dietary protein is affecting calcium absorption. Therefore, the purpose of this research is to evaluate whether dietary protein-induced changes in gastric acid secretion explain the observed changes in intestinal calcium absorption. We have compelling in vitro data that amino acids can stimulate gastric acid secretion. We have found that this occurs via allosteric activation of the calcium sensing receptor expressed on the gastric acid-secreting parietal cells. At a fixed concentration of extracellular calcium, addition of L but not D isomers of specific amino acids activates the calcium sensing receptor and stimulates parietal cell acid production. We hypothesize that dietary protein induced gastric acid production increases calcium solubility and bioavailability thereby increasing its absorption. We will test this hypothesis in humans by quantifying the impact of dietary protein on intestinal calcium absorption in subjects who cannot make gastric acid. We will measure intestinal calcium absorption in healthy adults as they consume either a high protein diet with concomitant administration of a proton pump inhibiting (PPI) drug or the same high protein diet with a placebo instead of a PPI. The order of the 2 interventions will be randomized, and study will be double-blind and placebo controlled. If our hypothesis is correct, then intestinal calcium absorption will be highest during the high protein diet with placebo, and lowest during the drug intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women age 18-45 years
* Caucasian or Asian descent due to increased risk of Osteoporosis

Exclusion Criteria:

* gastrointestinal diseases
* osteoporosis
* diabetes
* hypertension
* liver disease
* thyroid disorders
* kidney disease
* kidney stones
* cancer
* heart disease
* eating disorders
* obesity
* hypogonadism
* amenorrhea
* oligomenorrhea
* abnormal serum FSH or estradiol levels
* birth control medication or other hormone-altering medications
* pregnancy
* Lifestyle factors such as:

  * smoking
  * excessive exercise (although moderate exercise is allowed)
  * prescription medications known to influence vitamin D or calcium metabolism or gastric acid
  * excessive body weight change during the past 6 months
  * food allergies
  * unusual eating habits or medically prescribed diets

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Insogna, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Hospital Research Unit, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 healthy women and men enrolled
Pre-assignment Details: Participants received either Esomeprazole or placebo first and then crossed over to receive the other intervention with a minimum 2 week washout in-between.
Groups:
- Intervention Esomeprazole First/Placebo Second: In this group this group received the intervention first and then the placebo
- Intervention Placebo First/Esomeprazole Second: In this group this group received the placebo first and then the intervention
Period: Overall Study
Arm/Group | Intervention Esomeprazole First/Placebo Second | Intervention Placebo First/Esomeprazole Second
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive 20 mg twice daily of either placebo or esomeprazole first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Intestinal Calcium Absorption
Description: This is completed by measuring the amount of calcium absorbed by utilizing dual stable calcium isotopes. It was hypothesized that we would see a percent decrease as a result of the proton pump inhibitor. Previous published data indicated a decline in calcium absorption of 6.6 +/- 5.5% when gastric pH is blocked.
Time Frame: Day 5 of a high protein diet
Measure: Mean (Standard Error); unit: percentage of calcium absorption
Groups:
- Esomeprazole: Esomeprazoled administered twice daily in either first or second intervention period
- Placebo: Placebo administered twice daily in either first or second intervention
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 12 | 12
percentage of calcium absorption | 34.2 (2.4) | 31.5 (2.1)

2. Secondary Outcome: Gastric pH
Description: The American Heritage Dictionary defines pH as "a measure of the acidity or alkalinity of a solution, numerically equal to 7 for neutral solutions, increasing with increasing alkalinity and decreasing with increasing acidity. The pH scale commonly in use ranges from 0 to 14." The normal pH range for stomach acid is between 1.5 and 3.5.
Time Frame: Day 5 of a high protein diet
Measure: Mean (Standard Error); unit: units on a scale of pH
Groups:
- Esomeprazole Study Drug: Esomeprazole 20 mg twice daily given as either the first or second intervention
- Placebo: Placebo 20 mg twice a day given as either the first or second intervention.
Arm/Group | Esomeprazole Study Drug | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale of pH | 5.38 (0.13) | 2.70 (0.44)

ADVERSE EVENTS:
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes